CLINICAL TRIAL: NCT06858241
Title: Patient Intake At the 'MOvement and REhabilitation (MO.RE.)' Clinic: a Retrospective Observational Study on the Appropriateness of Access and the Needs Expressed by Patients. (BACKMORE2024)
Brief Title: Patient Intake At the 'MOvement and REhabilitation (MO.RE.)
Acronym: BACKMORE2024
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 299/2024/OSS/AUSLRE
Record Dates: First submitted 2025-02-04; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Oncologic Complications
Keywords: Onc-hematological patients; Physical Activity; Physical Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients who requested a consultation at the MO.RE. clinic between August 2022 and June 2024: Patients with a history of malignant tumor diagnosis, managed by the Oncology and Hematology Units that need a MO.RE. clinic consultation

SUMMARY:
In recent years, there has been an exponential increase in studies regarding the benefits of physical activity in oncology, with significant results on improving both physical and psychological outcomes. When appropriately dosed, physical activity can help individuals with a history of cancer to cope with pain and Cancer-Related Fatigue, and improve their quality of life, both during and after cancer treatments.

Given the incidence and prevalence of cancer, along with the increase in survival due to advancements in cancer care, it is becoming increasingly important to promote an active lifestyle.

For this reason, in August 2022, the MOvement and REhabilitation (MO.RE.) clinic was opened by the S.C. of MFR, dedicated to individuals with a history of cancer at any stage of treatment, with the aim of offering consultations with an experienced physiotherapist to personalize a physical activity program that can help regain a good quality of life, return to daily activities, and prevent the onset of other diseases and recurrences.

The clinic also provides therapeutic education activities, following WHO guidelines, on proper lifestyle for wellness and secondary prevention.

The aim of our study is to retrospectively analyze the patients who requested a consultation at the MO.RE. clinic between August 2022 and June 2024, in order to describe and evaluate the appropriateness of access to the clinic, the expressed needs, and some clinical and rehabilitative data."

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignant tumor
* Access to the MO.RE. clinic for recommendations on exercise/physical activity
* Age over 18 years

Exclusion Criteria:

* Language barrier
* Conditions that prevent the individual from performing physical activity independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of malignant tumor diagnosis, managed by the Oncology and Hematology Units of the USL-IRCCS of Reggio Emilia, who requested a consultation at the MO.RE. clinic between August 2022 and June 2024
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Number of cancer patients who accessed the MO.RE. service, matching appropriateness criteria | 2 years
  The referral of the patient is considered appropriate, if the patient corresponds to these criteria:
  * cancer patient needing information about a personalized physical activity program
  * patient with a good performance status evaluated according to ECOG performance status scale (score 0 or 1)
  * absence of bone metastases.

SECONDARY OUTCOMES:
Sample description by socio-demographic data | 2 years
  To describe the sample, data will be collected at the first access at MO.RE. service, concerning:
  * age (measured in years)
  * gender (M/F)
  * education level (number of years attending school)
  * occupation (descriptive)
  * Municipality of residence (distance from hospital).
Sample description by clinical data | 2 years
  To describe the sample, data will be collected at the first access at MO.RE. service, concerning:
  * Performance status at the first access to MO.RE. service
  * Location of primary tumor
  * Ongoing anticancer therapy
  * surgery (type of intervention and time elapsed between surgery and access to the MO.RE. service)
  * Complications, if any
  * Presence of bone metastases
  * Description of any ongoing or completed rehabilitation program
  * Amount of physical activity pre- and post-cancer diagnosis
  * Signs and symptoms related to cancer or anticancer therapies
  * patients specific needs
  * patient referral (how did patients access MO.RE. service? by oncologist referral, by other patients suggestion, information by social media, other)
Number of cancer patients who needed counselling on physical activity and self-managed exercise after MO.RE. access | 2 years
  At the end of the evaluation at MO.RE. service, a number of empowered cancer patients are able to self-manage physical activity in their life, after receiveing specific information about type, intensity, timing and frequency of appropriate exercise.
Number of cancer patients who needed counselling on physical activity and self-managed exercise after MO.RE. access | 2 years
  At the end of the evaluation at MO.RE. service, a number of cancer patients need a supervision by a physiotherapist, to become able to self-manage physical activity in their life. These patients receive a supervised rehabilitation program, to learn specific type, intensity, timing and frequency of appropriate exercise matching their condition.
Number of cancer patients who needed a physiatrist evaluation before exercise | 2 years
  At the end of the evaluation at MO.RE. service, a number of cancer patients need a physiatrist consultation, to avoid adverse events correlated with bone metastases or because they need a specific medical evaluation before exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Fugazzaro, MD, Principal Investigator — AUSL-IRCCS of Reggio Emilia
Locations (1):
- AUSL-IRCCS of Reggio EmiliaOperational Unit of Physical Medicine and Rehabilitation AUSL - IRCCS Reggio Emilia, Reggio Emilia, Emilia Romagna 42123, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No